CLINICAL TRIAL: NCT05939570
Title: Pediatric Day-of-Surgery Cancellations and the Association With Neighborhood Opportunity and Indices of Vulnerability : Phase II
Brief Title: DOSC and Association With Neighborhood Opportunity: Phase II
Status: Recruiting | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Brittany Willer, MD, Nationwide Children's Hospital
Other Study IDs: STUDY00003198
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Day of Surgery Cancellations
Keywords: Pediatrics; Day of Surgery Cancellations
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Interview — Prospective, semi-structured, qualitative interview.

SUMMARY:
Prospective, qualitative interview study to explore factors associated with pediatric day of surgery cancellations (DOSC) from the prospective of parents with hopes the interviews will reveal additional vulnerabilities not included in COI 2.0 that predispose to DOSC.

DETAILED DESCRIPTION:
We plan to prospectively study vulnerability factors that contribute to day of surgery cancellations (DOSC) by conducting a qualitative study using semi-structured interviews with families cancelled the day of surgery. We plan to enroll between 20-30 families using convenience sampling. Based on preliminary data, we anticipate that most families will come from minority racial and ethnic groups and parents of non-English primary language (NEPL) - these interviews will be conducted via an interpreter. Interviews will be structured to explore surgical care utilization themes based on the Gelberg-Anderson Behavioral Model for Vulnerable Populations including 1) Parental knowledge and attitudes regarding surgical services, 2) family and community resources, 3) Perceived surgical conditions and perceived need for surgical services, and 4) use of surgical services and difficulties accessing them. Family recruitment will be ongoing and will continue until we have reached saturation of themes. The data generated from this study will lay the foundation for a multi-layered intervention at the hospital level to allow patients to be triaged according to COI 2.0, race/ethnicity, NEPL status, and other vulnerabilities. This will enable adaptation of hospital pre-operative procedures (i.e. NPO preoperative calls) to reduce DOSC.

ELIGIBILITY:
Inclusion Criteria:

* Parents/guardians of children <18 who had a day of surgery cancellation
* Parents/guardians speak English, Spanish, Somali, Nepali or Arabic.

Exclusion Criteria:

* Parents/guardians speak a different language other than above listed.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Parents/guardians of children <18 who had a day of surgery cancellation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Factors associated with DOSC | Identified during interview.

SECONDARY OUTCOMES:
Additional vulnerabilities not included in COI 2.0 that predispose to DOSC | Identified during interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No